CLINICAL TRIAL: NCT04582734
Title: Screening and Intervention Reducing Anxiety in Patients With Cardiac Disease: The Heart & Mind Trial
Brief Title: Screening and Intervention Reducing Anxiety in Patients With Cardiac Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Herlev and Gentofte Hospital (Other); Aalborg University Hospital (Other); Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Selina Kikkenborg Berg, Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: The Heart & Mind Trial
Record Dates: First submitted 2020-09-24; First posted 2020-10-09 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Cognitive Therapy; Anxiety Disorders; Heart Diseases
Keywords: Cognitive Therapy; Anxiety; Heart diseases
MeSH Terms: conditions — Anxiety Disorders; Heart Diseases | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Masking Description: Because of the conditions required for psycho-educational interventions, it is not possible to blind the intervention staff and patients. All baseline information and clinical interviews are collected and performed before randomization. Physical tests, data collection, data management and administration will be done by blinded staff. Statistical analysis of outcomes and conclusions from these will be blinded. Results of the trial are analysed by an independent statistician, and the results will be interpreted by the research group. The conclusion will be prepared in two versions, before the allocation code is broken, with the two arms alternately assumed as intervention (one that assumes that arm A is the intervention, and second, that assumes that the arm B intervention).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group - cognitive behavioral therapy (Experimental): The intervention consists of three parts: 1) screening of hospitalised and outpatient cardiac patients at four university hospitals using the Hospital Anxiety and Depression Scale (HADS), scores ≥8 are invited to participate. (2) Assessment of type of anxiety by Structured Clinical Interview for DSM Disorders (SCID). (3) Investigator-initiated randomised clinical superiority trial with blinded outcome assessment, with 1:1 randomisation to cognitive-behavioural therapy (CBT) performed by a cardiac nurse with CBT training, plus usual care or usual care alone.The intervention is considered finalized if the patient has a HADS-A score under 8 two times in a row. The intervention group will receive usual care as well.
  Interventions: Behavioral: Cognitive-behavioural therapy
- Usual Care group (No Intervention): The usual care group (control group) will receive usual care which consists cardiac disease control and treatment.

INTERVENTIONS:
Behavioral: Cognitive-behavioural therapy — Cognitive-behavioural therapy intervention
  Arms: Intervention group - cognitive behavioral therapy

SUMMARY:
The hypothesis is that there is a significant difference in anxiety scores between intervention and usual care group after intervention. The aim of Heart & Mind Trial is (I) to determine the type of anxiety in cardiac patients and (ii) to investigate the effect of individual cognitive behavioural therapeutic intervention to reduce anxiety in patients with cardiac disease and anxiety compared to usual care.

DETAILED DESCRIPTION:
The Heart & Mind Trial is an investigator-initiated randomised clinical superiority trial with blinded outcome assessment, including four university hospitals, with 1:1 randomisation to cognitive therapy plus usual care or usual care alone.

The intervention: all patients receive usual care. Patients in the intervention group will receive an intervention based on cognitive behavioral therapy.

The intervention consists of three steps: (1) screening of hospitalised and outpatient cardiac patients at four university hospitals using the Hospital Anxiety and Depression Scale (HADS), scores ≥8 are invited to participate. (2) Assessment of type of anxiety by Structured Clinical Interview for DSM Disorders (SCID). (3) Investigator-initiated randomised clinical superiority trial with blinded outcome assessment, with 1:1 randomisation to cognitive-behavioural therapy (CBT) performed by a cardiac nurse with (CBT) training, plus usual care or usual care alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥18 years
* Diagnosed with cardiac disease
* Speak and understand Danish
* Score ≥8 on the Hospital Anxiety and Depression Scale - Anxiety (HADS-A)
* HADS-A score must exceed the HADS-D score
* Gives written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) Anxiety | 5 months
  Primary outcome is anxiety measured by HADS-A. HADS is a 14 item questionnaire that assesses anxiety and depression level in medical ill persons who are not admitted in psychiatric wards.
  Scores of 0 to 7 for either subscale are regarded as normal and scores of 8 to 10 suggest the presence of a mood disorder. Scores of 11 and above suggest probable presence of a mood disorder.

SECONDARY OUTCOMES:
Becks Anxiety Inventory (BAI) | Baseline, 5 months and 12 months
  Becks Anxiety Inventory is a brief self-reported measure of anxiety with a focus on somatic symptoms of anxiety and was developed as a measure to discriminate between anxiety and depression. Respondents indicated how much each symptom has bothered them during the past week on a 4-point Likert scale ranging from 0 (not at all) to 3 (severely).
  The BAI score ranges from 0-63.
Heart rate variability (HRV) | Baseline, 5 months
  HRV is measured using a Holter monitor. HRV are responsive to sympathetic activity, which can be increased by anxiety. HRV refers to the beat-to-beat variation in the RR interval and is a marker of autonomic nervous system activity.
Hospital Anxiety and Depression Scale (HADS) Anxiety | Baseline
  Primary outcome is anxiety measured by HADS-A. HADS is a 14 item questionnaire that assesses anxiety and depression level in medical ill persons who are not admitted in psychiatric wards.
  Scores of 0 to 7 for either subscale are regarded as normal and scores of 8 to 10 suggest the presence of a mood disorder. Scores of 11 and above suggest probable presence of a mood disorder.

OTHER OUTCOMES:
Cortisol level | Baseline, 5 months
  The level of Cortisol measured in a blood sample.
C-reactive protein (CRP) | Baseline, 5 months
  CRP is measured in a blood sample.
Heart Quality of Life (HeartQoL) | Baseline, 5 months and 12 months
  The questionnaire measures health-related quality of life in patients with ischemic heart disease, specifically angina, myocardial infarction or ischemic heart failure. The questionnaire consists of 14 items and provides two subscales; a 10-item physical subscale and a 4-item emotional subscale which each are scored from 0 to 3. The score ranges from 0-42. A higher score indicates a better heart related quality of life.
Health behaviour - Sleep quality | Baseline, 5 months and 12 months
  Patients' own evaluation of sleep quality.
Health behaviour - Physical activity | Baseline, 5 months and 12 months
  Patients' own evaluation of physical activity.
Health behaviour - Alcohol | Baseline, 5 months and 12 months
  Number of alcohol units per week.
Health behaviour - Smoking | Baseline, 5 months and 12 months
  Number of cigarettes per day.
Health behaviour - Weight. | Baseline, 5 months and 12 months
  Weight in kilogram.
Number of participants with admissions, readmissions and number of patients who died during the trial period. | 12 months
  Data regarding admissions, redadmissions and mortality through registers.
Hospital Anxiety and Depression Scale (HADS) Depression | Baseline, (intervention group: every CBT session), 5 months and 12 months
  Depression measured by HADS-D. HADS is a 14 item questionnaire that assesses anxiety and depression level in medical ill persons who are not admitted in psychiatric wards.
  Scores of 0 to 7 for either subscale are regarded as normal and scores of 8 to 10 suggest the presence of a mood disorder. Scores of 11 and above suggest probable presence of a mood disorder.
Hospital Anxiety and Depression Scale (HADS) Anxiety | 12 months
  Primary outcome is anxiety measured by HADS-A. HADS is a 14 item questionnaire that assesses anxiety and depression level in medical ill persons who are not admitted in psychiatric wards.
  Scores of 0 to 7 for either subscale are regarded as normal and scores of 8 to 10 suggest the presence of a mood disorder. Scores of 11 and above suggest probable presence of a mood disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Selina K Berg, PhD, Principal Investigator — Copenhagen University Hospital, Rigshospitalet, Denmark.
Locations (4):
- Denmark (4):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus N
  - Rigshospitalet, Copenhagen O
  - Herlev and Gentofte Hospital, Hellerup

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berg SK, Herning M, Schjodt I, Thorup CB, Juul C, Svendsen JH, Jorgensen MB, Risom SS, Christensen SW, Thygesen L, Rasmussen TB. The heart & mind trial: intervention with cognitive-behavioural therapy in patients with cardiac disease and anxiety: randomised controlled trial protocol. BMJ Open. 2021 Dec 3;11(12):e057085. doi: 10.1136/bmjopen-2021-057085. PMID 34862302